CLINICAL TRIAL: NCT07206082
Title: LUDICO Study: Effectiveness and Safety of Coronary Laser in UnDIlatable or unCrOssable Lesions
Brief Title: Coronary Laser in Undilatable or Uncrossable Lesions
Acronym: LUDICO
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Alfonso Jurado, MD, PhD, Principal investigator, Hospital Universitario La Paz
Other Study IDs: 5502
Record Dates: First submitted 2025-09-10; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Calcified Coronary Artery Disease; In Stent Restenosis; Chronic Total Occlusion (CTO)
Keywords: Percutaneous coronary intervention; excimer laser coronary atherectomy; intravascular imaging; optical coherence tomography; complex coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- undilatable lesions: expansion <80% of the distal vessel diameter after inflation of a 1:1 non-compliant balloon at 18 atm
  Interventions: Device: Laser atherectomy
- uncrossable coronary lesions: (not crossable after using a small-profile balloon with adequate support, according to operator´s discretion
  Interventions: Device: Laser atherectomy

INTERVENTIONS:
Device: Laser atherectomy — ELCA procedure will be performed using the Spectranetics CVX300 (Spectranetics, Colorado Spring, CO, USA) and the latest generation Philips Laser System Excimer (Philips, San Diego, CA, USA) System, which is based on pulsed xenon-chlorine laser catheters capable of delivering excimer energy (wavelength 308 nm, pulse length 185 ns) from 30 to 80 mJ/mm2 (fluencies) at pulse repetition rates from 25 to 80 Hz.
  The ELCA technique will be performed according to current recommendations (18). The laser probe size will be at the operator´s discretion among the available options (rapid exchange concentric 0.9 mm, 1.4 mm, 1.7mm or 2.0mm). The selection of fluence, and repetition rate will be left to the operator. A saline infusion technique will be recommended, although application of laser with blood or contrast will be recommended in resistant lesions. In the event of unsuccessful initial therapy, additional plaque modification techniques may be employed at the discretion of the operator and wi

SUMMARY:
This will be an investigator-initiated, multicentre, single-arm, open-label, prospective observational study. Patients with indication for PCI and undilatable (non-compliant balloon dilatation <80% at burst pressure) or uncrossable (not crossable with a "small-profile balloon" with adequate support, according to operator´s discretion) coronary lesions treated with ELCA will be included. Intravascular imaging will be highly recommendable and analysed in a central core-laboratory. Device success, angiographical success, procedural success, clinical success and related complications will be evaluated. Patients will be followed for 1 year after the procedure and clinical events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years.
* Patients with either stable coronary artery disease or acute coronary syndromes as the clinical presentation.
* Patients with severe coronary lesions (>70% by visual estimation) in native vessels or coronary bypass grafts.
* "Uncrossable" coronary lesions (i.e., lesions that cannot be crossed with a 0.7:1 balloon after successful guidewire passage) or "Undilatable" lesions (i.e., those in which balloon dilation with a 1:1 non-compliant balloon at 18 atm results in less than 80% expansion relative to the distal reference vessel diameter; this group includes both de novo lesions and in-stent restenosis or underexpanded stents).

Exclusion Criteria:

* Patients with known allergies to aspirin (ASA), clopidogrel, prasugrel, or ticagrelor.
* Patients unable to provide informed consent, either personally or through a legal representative.
* Patients with clinical or hemodynamic instability defined as: sustained hypotension (systolic blood pressure ≤ 90 mmHg for ≥ 30 minutes or use of pharmacological and/or mechanical support to maintain an SBP ≥90 mmHg) or evidence of end-organ hypoperfusion including urine output of <30 mL/h, cool extremities, altered mental status, and/or serum lactate >2.0 mmol/L.
* Patients with significant comorbidities and a life expectancy of less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for PCI and undilatable or uncrossable lesions treated with ELCA
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Laser Success | From enrollment to the end of the procedure at 4 hours.
  For uncrossable lesions, it will be defined as the ability of the laser catheter to cross the lesion. Laser success will be also considered in cases in which the laser catheter cannot cross the lesion but its application proximal to it allows subsequent crossing of balloons. For undilatable lesions, laser success will be defined as successful balloon dilation (sized 1:1 to the vessel diameter), with adequate expansion (>80% in two orthogonal projections) following laser therapy without the need of other plaque modification technique.

SECONDARY OUTCOMES:
Angiographic success | From enrollment to the end of the procedure at 4 hours.
  Thrombolysis in myocardial infarction (TIMI) 3 final flow and a diameter stenosis <20%.
Procedural success | From enrollment to the end of the procedure at 4 hours.
  Angiographic success without severe procedural complications (death, coronary perforation, abrupt vessel closure, flow-limiting dissection).
Intracoronary imaging-based success | From enrollment to the end of the procedure at 4 hours.
  Stent expansion ≥80% [OCT or intravascular ultrasound (IVUS)] or a minimal stent area (MSA) ≥4.5mm2 in OCT or ≥5.5mm2 in IVUS.
Events at 1 year | From enrollment to 1 year after the procedure
  Clinical events and antiplatelet therapy will be recorded, including the rate of major cardiovascular events (MACE), defined as the occurrence of cardiac death, target vessel acute myocardial infarction (MI), target vessel revascularization (TVR), and stent thrombosis), death, cardiovascular death, non-fatal MI, target lesion revascularization (TLR), TVR, stroke and bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be publicly shared; however, data sharing may be considered in selected cases upon reasonable request and with sufficient justification.